CLINICAL TRIAL: NCT03051282
Title: Genetic Determinants of ACEI Prodrug Activation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Haojie Zhu, Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HUM00114879
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Enalapril; Enalaprilat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- non-carrier control group (Active Comparator): Subjects who do not carry the CES1 variant G143E (rs71647871) will receive 10 mg Enalapril orally once daily for 7 consecutive days.
  Interventions: Drug: Enalapril
- G143E carriers group (Active Comparator): Subjects who carry the CES1 variant G143E (rs71647871) will receive 10 mg Enalapril orally once daily for 7 consecutive days.
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Enalapril — Study participants in both arms will be treated with 10 mg enalapril orally once daily for seven consecutive days
  Other Names: Vasotec®

SUMMARY:
Angiotensin-converting enzyme inhibitors (ACEIs) are among the most frequently prescribed medications worldwide for the treatment of essential hypertension, left ventricular systolic dysfunction, acute myocardial infarction, and prevention of the progression of diabetic nephropathy. However, the outcome of ACEI treatment varies significantly between individuals and selected populations. Suboptimal response, therapeutic failure, and significant side effects are commonly documented in patients receiving ACEI therapy. Approximately 80% of the ACEIs available for use in the US are synthesized as esterified prodrugs in order to improve otherwise poor oral bioavailability of the active molecule. The activation of ACEI prodrugs primarily occurs in the liver via metabolic de-esterification of the parent drug. The critical activation step is essential in delivering a successful therapeutic outcome since the active metabolites are approximately 10-1000 times more potent relative to their respective parent compounds. Carboxylesterase 1 (CES1), the most abundant hydrolase in the liver, is responsible for the activation of ACEI prodrugs in humans. Marked interindividual variability in CES1 expression and activity has been documented, which results in varied therapeutic efficacy and tolerability of many drugs serving as substrates of CES1. Genetic variation of CES1 is considered to be a major factor contributing to variability in CES1 function. The study team proposes to conduct a multiple-dose healthy volunteer study to evaluate the impact of CES1 genetic variation on the activation, pharmacokinetics, and pharmacodynamics of enalapril, a model ACEI prodrug activated by CES1. The completion of this study will represent a major step towards the establishment of an evidence base from which a more individualized use of ACEI prodrugs can emerge.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be male and female (50:50) between the ages of 18-55 years
* Females must have a negative urine pregnancy test prior to the study
* All subjects must have no clinically significant diseases or clinically significant abnormal laboratory values as assessed during the screening medical history, nursing assessment, and laboratory evaluations
* Informed consent must be signed by the eligible subject prior to the initiation of any study procedures

Exclusion Criteria:

* The presence of a known medical condition that would preclude the use of enalapril
* The presence of any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion.
* A positive urine pregnancy test in the MCRU prior to the study
* No subjects weighing under 50 kg will be selected
* The lack of use of acceptable methods of birth control unless abstinent
* Subjects who regularly take medications, vitamins, herbal supplements
* The use of any illicit drugs or habitual consumption of large quantities of ethanol (>3 drinks/day)
* The consumption of grapefruit or grapefruit juice a week prior to, and during the study
* Asians will not be included in the study as the CES1 SNP G143E is absent in this population
* Subjects hypersensitive to enalapril
* Subject with a history of angioedema
* Smokers

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The measurements of the mean area under the curve (AUC) of enalaprilat plasma concentrations | 72 hours
  To compare the mean AUC of enalaprilat plasma concentrations between the non-carrier control and the G143E carriers groups

SECONDARY OUTCOMES:
The measurements of the maximum enalaprilat plasma concentrations | 72 hours
  To compare the maximum enalaprilat plasma concentrations between the non-carrier control and the G143E carriers groupsG143E carriers groups
The measurements of angiotensin converting enzyme (ACE) activity in plasma | 72 hours
  To compare the plasma ACE activity between the non-carrier control and the G143E carriers groupsG143E carriers groups following enalapril treatment
The measurements of blood pressures (BPs) following enalapril treatment | 72 hours
  To compare the changes of BPs between the non-carrier control and the G143E carriers groupsG143E carriers groups following enalapril treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Her LH, Wang X, Shi J, Choi HJ, Jung SM, Smith LS, Wu AH, Bleske BE, Zhu HJ. Effect of CES1 genetic variation on enalapril steady-state pharmacokinetics and pharmacodynamics in healthy subjects. Br J Clin Pharmacol. 2021 Dec;87(12):4691-4700. doi: 10.1111/bcp.14888. Epub 2021 May 26. PMID 33963573